CLINICAL TRIAL: NCT05898555
Title: Validation of Smart Garments for Gait and Balance Assessment
Brief Title: Validation of Smart Garments for Gait Classification
Status: Recruiting | Type: Observational
Sponsor: Myant Medical Corp. (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: Myant/Waterloo/42689
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Gait analysis; Wearable electronic devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Gait study protocol
  Interventions: Device: Skiin garment and pods

INTERVENTIONS:
Device: Skiin garment and pods — Participants will be asked to wear a Skiin smart garment over their own clothes.
  Small motion capture markers will be placed on their body and pressure-sensitive insoles placed into their shoes to measure the pressure underneath their feet during the study tasks.
  Once the sensors are ready for collection, participants will be asked to complete 5 tasks associated with their daily activities: 1. Locomotion; 2. Lower limb strength - repeated sit-to-stand-to-sit transitions; 3. Lower limb strength and locomotion - Timed Up and Go; 4. Free walking during a 2min walk; 5. Standing balance, postural control.

SUMMARY:
The aim of this study is therefore to validate Myant SKIIN garments for the purpose of gait and balance assessment. To achieve this, we recruit young healthy adults from the University of Waterloo to wear Skiin products (see Fig. 1). Participants will be asked to perform a number of scripted gait and balance tasks.

DETAILED DESCRIPTION:
Specific objectives of this study are:

1. To validate Skiin gait characterization algorithm (based on single garment solutions - already developed based on a literature and a previous study conducted at the University of Waterloo);
2. To develop algorithms for multi-garments solutions that aim to extract additional kinematic parameters such as joint angles.

Gait metrics from Skiin garments will be compared to metrics from a gold standard measurement (Vicon motion capture) to indicate accuracy, precision and reliability.

ELIGIBILITY:
Inclusion Criteria:

- Healthy male and female adults aged 18y - 64y old

Exclusion Criteria:

- Self-reported lower limb conditions, neurological disorders, history of concussion/brain trauma, and/or condition limiting exercise is to mitigate additional risk for injury and/or adverse reactions associated with exercise.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience-sample of 20 healthy individuals will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Error in step length metric | Collection during the single study session of 1.5 hours.
  The difference between step lengths calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in stride length metric | Collection during the single study session of 1.5 hours.
  The difference between stride length calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in cadence metric | Collection during the single study session of 1.5 hours.
  The difference between cadence calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in step duration (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between step duration (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in stride duration (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between stride duration (s), and its asymmetry calculated from Skiin data for each scripted gait tasks.
Error in stance duration (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between stance duration (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in swing duration (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between swing duration(s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in initial double support (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between double support (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in terminal double support (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between terminal double support (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in double support (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between double support (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in single limb support (s) metric, and its asymmetry | Collection during the single study session of 1.5 hours.
  The difference between single limb support (s), and its asymmetry calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in gait speed metric | Collection during the single study session of 1.5 hours.
  The difference between gait speed calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in stride speed metric | Collection during the single study session of 1.5 hours.
  The difference between stride speed calculated from Skiin data and from Vicon data for each scripted gait tasks.
Error in mean CoM sway distance | Collection during the single study session of 1.5 hours.
  The difference between sway distance of the Center of mass calculated from Skiin data and from Vicon data for each scripted balance tasks.
Error in mean CoM sway velocity | Collection during the single study session of 1.5 hours.
  The difference between sway velocity of the Center of mass calculated from Skiin data and from Vicon data for each scripted balance tasks.
Error in CoM sway area | Collection during the single study session of 1.5 hours.
  The difference between sway area of the Center of mass calculated from Skiin data and from Vicon data for each scripted balance tasks.
Error in CoM sway frequency | Collection during the single study session of 1.5 hours.
  The difference between sway frequency of the Center of mass calculated from Skiin data and from Vicon data for each scripted balance tasks.

CONTACTS AND LOCATIONS:
Overall Officials: James Tung, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo - Engineering 7, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided